CLINICAL TRIAL: NCT00283244
Title: Randomized Phase II Study of First-Line Treatment With Gemcitabine vs. Erlotinib vs. Gemcitabine and Erlotinib in Elderly Patients With Stage IIIB/IV Non-Small Cell Lung Cancer
Brief Title: Ph II Gemcitabine, Erlotinib, and Gemcitabine With Erlotinib/Elderly Patients W/ IIIB/IV NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 0512; P30CA016086 (NIH); UNC-LCCC-0512 (Other: UNC IRB #05-2256)
Record Dates: First submitted 2006-01-24; First posted 2006-01-27 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Lung Cancer
Keywords: stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A (Active Comparator): Patients receive gemcitabine hydrochloride 1200mg/m2 IV on days 1 and 8. Patients with progressive disease may cross over to arm B.
  Interventions: Drug: gemcitabine hydrochloride
- Arm B (Experimental): Patients receive oral erlotinib hydrochloride 150mg p.o. daily on days 1-21.
  Interventions: Drug: erlotinib hydrochloride
- Arm C (Experimental): Patients receive gemcitabine hydrochloride 1000mg/m2 IV on days 1 and 8 and erlotinib hydrochloride 100mg p.o. daily
  Interventions: Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Drug: erlotinib hydrochloride — given orally
  Other Names: Tarceva
  Arms: Arm B; Arm C
Drug: gemcitabine hydrochloride — given IV
  Other Names: Gemzar
  Arms: Arm A; Arm C

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. It is not yet known whether gemcitabine and erlotinib are more effective when given alone or together in treating non-small cell lung cancer.

PURPOSE: This randomized phase II trial is studying gemcitabine and erlotinib to compare how well they work when given alone or together as first-line therapy in treating older patients with stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Compare the progression-free survival rate of older patients with stage IIIB or IV non-small cell lung cancer treated with gemcitabine hydrochloride vs erlotinib hydrochloride vs gemcitabine hydrochloride and erlotinib hydrochloride as first-line therapy.

Secondary

* Determine the response rate in patients receiving these regimens.
* Determine the overall survival rate in patients receiving these regimens.
* Determine the toxicity profile of these regimens in these patients.
* Determine the quality of life of patients receiving these regimens.

OUTLINE: This is a randomized, open-label, controlled, parallel group, multicenter study. Patients are stratified by gender, smoking status (never or light vs current or former), and ECOG performance status (0-1 vs 2). Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive gemcitabine hydrochloride IV on days 1 and 8. Patients with progressive disease may cross over to arm II.
* Arm II: Patients receive oral erlotinib hydrochloride daily on days 1-21.
* Arm III: Patients receive gemcitabine hydrochloride as in arm I and erlotinib hydrochloride as in arm II.

In all arms, treatment repeats every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed every 2 months for 3 years.

ELIGIBILITY:
Inclusion Criteria Histologic or cytologic diagnosis of stage NSCLC ECOG Performance Status (PS) 0-2 Absolute Neutrophil Count (ANC) ≥ 1.5 Platelets ≥ 100,000 Hemoglobin ≥ 8.0 g/dl Aspartate aminotransferase (AST)/Alanine aminotransferase (ALT) ≤ 2.5 upper limit of institutional normal (ULN) Alkaline phosphatase ≤ 4 x ULN Total Bilirubin below or equal to upper institutional normal limits Serum Creatinine ≤ 1.5 x ULN Patients may have received 1 prior treatment in the adjuvant setting, but time since prior chemotherapy must be ≥1 year. Although the protocol specifically says adjuvant therapy, we believe neoadjuvant is similar and patients who have received neo-adjuvant (pre-operative) rather than classic adjuvant (post-operative) therapy are similar and should not be distinguished. Therefore, patients may have received

1 prior treatment in the neo-adjuvant setting as well. Treated brain metastases are eligible provided the patient is asymptomatic and meets the above criteria, including PS. Measurable disease by RECIST criteria Ability to give informed consent

Exclusion Criteria Patients with a history of severe hypersensitivity to gemcitabine. Incompletely healed from previous oncologic or other major surgery. Pregnancy or breast feeding (women of childbearing potential are not expected to be enrolled in this study given minimum age) Patients with severe co-morbid illness. Patients unable to participate in the QOL assessments.

Ages: 70 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-03; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas E Stinchcombe, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (11):
- United States (11):
  - Highlands Oncology Group - Fayetteville, Fayetteville, Arkansas
  - Summit Cancer Care, Savannah, Georgia
  - Evanston Hospital, Evanston, Illinois
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Batte Cancer Center at Northeast Medical Center, Concord, North Carolina
  - Cape Fear Valley Medical Center Cancer Center, Fayetteville, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Kingsport Hematology-Oncology Associates, Kingsport, Tennessee
  - University of Tennessee Cancer Institute - Memphis, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No
There is no plan to share any individual participant data.

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://clinicaltrials.gov/ct2/show/NCT00283244

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited for this study between March 2006 and May 2010
Pre-assignment Details: Of the 160 patients who signed informed consent, 13 didn't start treatment for the following reasons: withdrew informed consent (5), referred to hospice (4), ineligible (3), and death before treatment (1). A patient received treatment on trial, but was determined to be ineligible due to incorrect diagnosis, and was thus not included in results.
Groups:
- Arm A (Gemcitabine): Patients receive gemcitabine hydrochloride 1200mg/m2 IV on days 1 and 8. Patients with progressive disease may cross over to arm B.
- Arm B (Erlotinib): Patients receive oral erlotinib hydrochloride 150mg p.o. daily on days 1-21.
- Arm C (Gemcitabine + Erlotinib): Patients receive gemcitabine hydrochloride 1000mg/m2 IV on days 1 and 8 and erlotinib hydrochloride 100mg p.o. daily
Period: Overall Study
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
Started | 44 | 51 | 51
Completed | 26 (19 patients went on to receive second line Erlotinib) | 0 (Patients treated until progression or unacceptable toxicity; 12 patients received 2nd line therapy) | 0 (Patients treated until progression or unacceptable toxicity; 9 patients received 2nd line therapy)
Not Completed | 18 | 51 | 51
Not completed — Adverse Event | 0 | 8 | 11
Not completed — Death | 4 | 3 | 2
Not completed — Lack of Efficacy | 8 | 32 | 26
Not completed — Withdrawal by Subject | 1 | 2 | 2
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Medical illness (other complicating dz) | 4 | 3 | 6
Not completed — Clinical deterioration | 1 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib) | Total
Number analyzed (Participants) | 44 | 51 | 51 | 146
Age, Continuous [Median (Full Range); unit: years] | 74 [70 to 86] | 76 [69 to 86] | 78 [70 to 90] | 76 [69 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 27 | 24 | 73
  Male | 22 | 24 | 27 | 73
Region of Enrollment [Number; unit: participants]
  United States | 44 | 51 | 51 | 146
Cancer Stage (TNM) [Number; unit: participants] — Anatomic stage for NSCLC is the American Joint Committee on Cancer (AJCC) TNM system, which is based on:
  Size of primary tumor (T) and whether it has grown into nearby areas. Spread to regional lymph nodes (N). Spread (metastasis; M) to other organs of the body. Once the T, N, and M categories have been determined, this information is combined into a prognostic group. Higher numbers (Roman numerals) mean the cancer is more advanced.
  participants
    IIIB (Any T, N3, M0 or T4, N2, M0) | 11 | 5 | 10 | 26
    IV (Any T, any N, M1a or M1b) | 33 | 46 | 41 | 120
ECOG Performance Status [Number; unit: participants] — A scale from 0-5 to describe a patient's level of functioning in terms of selfcare ability and activity level.
  0, Fully active
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  participants
    0 | 10 | 7 | 6 | 23
    1 | 21 | 29 | 29 | 79
    2 | 13 | 14 | 14 | 41
    Missing at baseline | 0 | 1 | 2 | 3
Smoking history [Number; unit: participants]
  Never or light smoker | 4 | 6 | 5 | 15
  Current or former smoker | 35 | 43 | 42 | 120
  Missing | 5 | 2 | 4 | 11
Histology [Number; unit: participants]
  Adenocarcinoma | 28 | 34 | 31 | 93
  Squamous | 7 | 5 | 8 | 20
  Large cell carcinoma | 1 | 0 | 0 | 1
  Not otherwise specified | 8 | 12 | 12 | 32
Cumulative Illness Rating scale for Geriatrics (CIRS-G) [Median (Full Range); unit: units on a scale] — A measure of co-morbidity burden rating the severity of chronic diseases in 14 individual body systems.
  Severity ratings:
  0=No problems.
  1. Current mild or past significant problem.
  2. Moderate disability or morbidity and/or requires first line therapy.
  3. Severe problem; constant, significant disability and/or hard to control chronic problems.
  4. Extremely severe problem; immediate treatment required; organ failure and/or severe functional impairment.
  Total score is a sum of the 14 item scores and may vary from 0 to 56. A higher score represents higher co-morbidity (worse health).
  units on a scale | 11.5 [0 to 25] | 10 [2 to 24] | 11 [4 to 24] | 11 [0 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: We would consider the combination of gemcitabine plus erlotinib or single agent erlotinib to be worthy of further study if there was an increased progressed-free survival. We would use an increase to 45% progression-free survival at 6 months as significant. Progression is defined using Response Evaluation Criteria in Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Six months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
Number analyzed (Participants) | 44 | 51 | 51
months | 3.7 [2.3 to 4.7] | 2.8 [1.4 to 3.4] | 4.1 [2.4 to 5]

2. Secondary Outcome: Response Rate
Description: The best overall response (BOR) is the best response recorded from the start of the treatment until disease progression-recurrence (taking as reference for progressive disease the smallest measurement recorded since the treatment started. The response rate was defined as the percentage of patients achieving a BOR of complete response or partial response. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Six months
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
Number analyzed (Participants) | 44 | 51 | 51
percentage of participants | 7 | 0 | 21

3. Secondary Outcome: Overall Survival
Description: Survival calculated from start of treatment to death from any cause for up to three years.
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
Number analyzed (Participants) | 44 | 51 | 51
Months | 6.8 [4.8 to 8.5] | 5.8 [3.0 to 8.3] | 5.6 [3.5 to 8.4]

4. Secondary Outcome: Toxicity
Description: Assessments for treatment toxicity will be done with each cycle according to CTCAE v3. Results listed here are grade >=3, treatment related hematologic events (all) and Grade>=3 treatment related non hematologic events that occurred in >=5% of patients in any arm. Adverse events (toxicities) are graded on a 5 point scale from 1 (mild) to 5 (lethal), with grades 3 and higher being severe or life threatening.
Time Frame: After each cycle/3 weeks, up to 3 years
Measure: Number; unit: participants
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
Number analyzed (Participants) | 44 | 51 | 51
participants
  Anemia (Grade>=3; treatment related) | 1 | 0 | 4
  Neutropenia (Grade>=3; treatment related) | 4 | 1 | 1
  Thrombocyopenia (Grade>=3; treatment related) | 3 | 1 | 2
  Dehydration (Grade>=3; treatment related) | 0 | 3 | 2
  Diarrhea (Grade>=3; treatment related) | 0 | 3 | 3
  Dyspnea (Grade>=3; treatment related) | 2 | 0 | 3
  Fatigue (Grade>=3; treatment related) | 4 | 1 | 5
  Rash (Grade>=3; treatment related) | 1 | 2 | 3

5. Secondary Outcome: Quality of Life (QOL)- Functional Assessment of Cancer Therapy for Lung Cancer (FACT-L) Trial Outcome Index-L (TOI-L)
Description: The FACT-L is the FACT-G and a lung cancer specific (LCS) subscale given at baseline, after each cycle and at end of treatment. The FACT-G is a 27 item measure of general QOL assessing function in 4 domains: physical well-being (PWB), social-family well-being (SFWB), emotional well-being (EWB) and functional well-being (FWB). Items are rated by patients on a Likert scale from 0 to 4. Higher scores represent better QOL. The TOI-L sums the PWB, FWB, and LCS subscale scores.
  A best response for TOI-L scores is based on change from baseline and coded as:
  a change >=+6 "improved", <= -6 "worsened" and otherwise "no change".
  A best overall score response is coded as:
  Improved (2 visit resp. of "improved" a min. of 28 days apart w/ no interim "worsened") No change (not "improved;" 2 visit resp. of "no change" or "improved" a min. of 28 days apart w/ no interim "worsened") Worsened (not "improved" or "no change;" 2 consecutive "worsened") Other (none of the above)
Time Frame: After each cycle/3 weeks
Measure: Number; unit: participants
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
Number analyzed (Participants) | 44 | 51 | 51
participants
  Improved | 5 | 6 | 7
  No change | 12 | 9 | 9
  Worsened | 11 | 12 | 9
  Other | 16 | 24 | 26

ADVERSE EVENTS:
Time Frame: Adverse events were followed for 30 days after cessation of treatment
Arm/Group | Arm A (Gemcitabine) | Arm B (Erlotinib) | Arm C (Gemcitabine + Erlotinib)
All-Cause Mortality (participants affected / at risk) | 1/44 | 3/51 | 3/51
Serious Adverse Events (participants affected / at risk) | 16/44 | 17/51 | 26/51
Other Adverse Events (participants affected / at risk) | 40/44 | 46/51 | 48/51
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Gemcitabine) (N=44) | Arm B (Erlotinib) (N=51) | Arm C (Gemcitabine + Erlotinib) (N=51)
Edema: Limb (Blood and lymphatic system disorders) | 0 | 1 (1) | 0
Hemoglobin (Blood and lymphatic system disorders) | 0 | 1 (1) | 2 (3)
Leukocytes (Total Wbc) (Blood and lymphatic system disorders) | 0 | 1 (1) | 0
Neutrophils/Granulocytes (Anc/Agc) (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0
Platelets (Blood and lymphatic system disorders) | 0 | 1 (1) | 1 (1)
Cardiac Ischemia/Infarction (Cardiac disorders) | 2 (2) | 0 | 1 (1)
Cardiac Troponin I (Ctni) (Cardiac disorders) | 1 (1) | 0 | 0
Cardiopulmonary Arrest, Cause Unknown (Non-Fatal) (Cardiac disorders) | 0 | 0 | 1 (1)
Hypotension (Cardiac disorders) | 0 | 0 | 2 (2)
Supraventricular And Nodal Arrhythmia - Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 1 (2)
Supraventricular And Nodal Arrhythmia - Sinus Tachycardia (Cardiac disorders) | 0 | 1 (1) | 0
Constipation (Gastrointestinal disorders) | 1 (1) | 0 | 0
Dehydration (Gastrointestinal disorders) | 0 | 3 (3) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 1 (1)
Hemorrhage, Gi - Abdomen Nos (Gastrointestinal disorders) | 0 | 0 | 2 (2)
Hemorrhage, Gi - Colon (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Hemorrhage, Gi - Jejunum (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Hemorrhage, Gi - Upper Gi Nos (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 3 (3)
Perforation, Gi - Colon (Gastrointestinal disorders) | 1 (1) | 0 | 0
Perforation, Gi - Small Bowel Nos (Gastrointestinal disorders) | 0 | 0 | 1 (1)
Trismus (Difficulty, Restriction Or Pain When Opening Mouth) (Gastrointestinal disorders) | 0 | 1 (1) | 0
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1)
Death Not Associated With Ctcae Term - Death Nos (General disorders) | 0 | 0 | 2 (2)
Death Not Associated With Ctcae Term - Multi-Organ Failure (General disorders) | 0 | 1 (1) | 0
Death Not Associated With Ctcae Term - Sudden Death (General disorders) | 1 (1) | 0 | 1 (1)
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 1 (1) | 1 (1) | 5 (5)
Fever (In The Absence Of Neutropenia, Where Neutropenia Is Defined As (General disorders) | 0 | 0 | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 | 0
Pancreatitis (Hepatobiliary disorders) | 0 | 1 (1) | 0
Autoimmune Reaction (Immune system disorders) | 1 (1) | 0 | 0
Colitis, Infectious (E.G., Clostridium Difficile) (Infections and infestations) | 1 (1) | 0 | 1 (2)
Infection (Documented Clinically Or Microbiologically) With Grade 3 Or (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils - Catheter-Relat (Infections and infestations) | 1 (1) | 0 | 0
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils - Lung (Pneumoni (Infections and infestations) | 1 (1) | 0 | 1 (1)
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils - Skin (Cellulit (Infections and infestations) | 1 (1) | 0 | 0
Creatinine (Investigations) | 0 | 1 (1) | 0
Sodium, Serum-Low (Hyponatremia) (Investigations) | 0 | 2 (2) | 0
Alkaline Phosphatase (Metabolism and nutrition disorders) | 0 | 1 (1) | 0
Ataxia (Incoordination) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 | 0
Muscle Weakness, Generalized Or Specific Area (Not Due To Neuropathy) (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Below knee amputation (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1)
Cns Cerebrovascular Ischemia (Nervous system disorders) | 1 (1) | 0 | 2 (2)
Dizziness (Nervous system disorders) | 0 | 0 | 1 (1)
Neuropathy: Motor (Nervous system disorders) | 0 | 0 | 1 (1)
Seizure (Nervous system disorders) | 0 | 1 (1) | 0
Speech Impairment (E.G., Dysphasia Or Aphasia) (Nervous system disorders) | 0 | 0 | 1 (1)
Syncope (Fainting) (Nervous system disorders) | 0 | 0 | 1 (1)
Confusion (Psychiatric disorders) | 1 (1) | 0 | 0
Mental Status (Psychiatric disorders) | 0 | 0 | 1 (2)
Psychosis (Hallucinations/Delusions) (Psychiatric disorders) | 0 | 0 | 1 (1)
Somnolence/Depressed Level Of Consciousness (Psychiatric disorders) | 1 (1) | 0 | 1 (1)
Hemorrhage, Gu - Retroperitoneum (Renal and urinary disorders) | 0 | 1 (1) | 0
Renal Failure (Renal and urinary disorders) | 0 | 3 (3) | 0
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 3 (3) | 10 (11)
Hemorrhage, Pulmonary/Upper Respiratory - Respiratory Tract Nos (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 1 (1)
Pain - Abdomen Nos (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 0
Pain - Chest/Thorax Nos (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0
Pleural Effusion (Non-Malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 | 2 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (2) | 1 (1)
Pulmonary Fibrosis (Radiographic Changes) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2)
Hypoxic Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2)
Rash: Acne/Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
Rash: Dermatitis Associated With Radiation - Chemoradiation (Skin and subcutaneous tissue disorders) | 0 | 1 (1) | 0
Inr (International Normalized Ratio Of Prothrombin Time) (Vascular disorders) | 0 | 0 | 1 (1)
Peripheal Arterial Ischemia (Vascular disorders) | 0 | 0 | 2 (2)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 3 (3) | 0 | 1 (1)
Post Obstructive Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Gemcitabine) (N=44) | Arm B (Erlotinib) (N=51) | Arm C (Gemcitabine + Erlotinib) (N=51)
Albumin, Serum-Low (Hypoalbuminemia) (Metabolism and nutrition disorders) | 2 (2) | 1 (3) | 3 (10)
Allergic Reaction/Hypersensitivity (Including Drug Fever) (Immune system disorders) | 2 (2) | 1 (1) | 0 (0)
Alt, Sgpt (Serum Glutamic Pyruvic Transaminase) (Investigations) | 0 (0) | 0 (0) | 3 (4)
Anorexia (Metabolism and nutrition disorders) | 13 (17) | 13 (15) | 16 (25)
Bilirubin (Hyperbilirubinemia) (Investigations) | 0 (0) | 2 (4) | 4 (6)
Cataract (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 3 (3) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 13 (16) | 8 (9) | 15 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (31) | 10 (11) | 5 (11)
Creatinine (Investigations) | 1 (1) | 3 (3) | 5 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 4 (5) | 6 (7)
Diarrhea (Gastrointestinal disorders) | 10 (17) | 26 (47) | 22 (37)
Dizziness (Nervous system disorders) | 10 (23) | 5 (7) | 6 (7)
Dry Skin (Skin and subcutaneous tissue disorders) | 3 (5) | 6 (6) | 3 (3)
Dyspnea (Shortness Of Breath) (Respiratory, thoracic and mediastinal disorders) | 17 (32) | 11 (13) | 15 (30)
Edema: Limb (General disorders) | 4 (4) | 8 (10) | 8 (9)
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 27 (46) | 23 (32) | 27 (49)
Fever (In The Absence Of Neutropenia, Where Neutropenia Is Defined As (General disorders) | 5 (7) | 2 (2) | 2 (2)
Glucose, Serum-High (Hyperglycemia) (Metabolism and nutrition disorders) | 6 (7) | 3 (3) | 6 (13)
Hearing (without monitoring program) (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 2 (2)
Heartburn/Dyspepsia (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1)
Hemoglobin (Investigations) | 17 (24) | 13 (21) | 24 (43)
Hemorrhage, Gi - Rectum (Gastrointestinal disorders) | 0 (0) | 3 (3) | 3 (3)
Hemorrhage, Pulmonary/Upper Respiratory - Bronchopulmonary Nos (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1) | 0 (0)
Hemorrhage, Pulmonary/Upper Respiratory - Nose (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1)
Hypotension (Vascular disorders) | 3 (3) | 4 (5) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2)
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils - Bronchus (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Injection Site Reaction/Extravasation Changes (Immune system disorders) | 2 (4) | 0 (0) | 1 (7)
Insomnia (Psychiatric disorders) | 3 (4) | 6 (6) | 6 (6)
Leukocytes (Total Wbc) (Investigations) | 6 (17) | 0 (0) | 3 (4)
Mood Alteration - Anxiety (Psychiatric disorders) | 4 (4) | 3 (3) | 3 (5)
Mood Alteration - Depression (Psychiatric disorders) | 1 (1) | 3 (6) | 2 (2)
Mucositis/Stomatitis (Clinical Exam) - Oral Cavity (Gastrointestinal disorders) | 1 (4) | 5 (7) | 7 (8)
Mucositis/Stomatitis (Functional/Symptomatic) - Oral Cavity (Gastrointestinal disorders) | 3 (3) | 1 (1) | 1 (1)
Muscle Weakness, Generalized Or Specific Area (Not Due To Neuropathy) (Musculoskeletal and connective tissue disorders) | 7 (7) | 2 (3) | 4 (5)
Nausea (Gastrointestinal disorders) | 9 (32) | 9 (11) | 16 (30)
Neuropathy: Sensory (Nervous system disorders) | 4 (5) | 0 (0) | 2 (3)
Neutrophils/Granulocytes (Anc/Agc) (Investigations) | 8 (16) | 0 (0) | 3 (3)
Ocular/Visual - Other (Specify, __) (Eye disorders) | 2 (2) | 0 (0) | 0 (0)
Pain - Abdomen Nos (Musculoskeletal and connective tissue disorders) | 4 (5) | 2 (2) | 6 (9)
Pain - Back (Musculoskeletal and connective tissue disorders) | 8 (15) | 3 (5) | 4 (6)
Pain - Bone (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Pain - Cardiac/Heart (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Pain - Chest Wall (Musculoskeletal and connective tissue disorders) | 4 (7) | 1 (1) | 4 (4)
Pain - Chest/Thorax Nos (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 3 (5)
Pain - Extremity-Limb (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 3 (10)
Pain - Head/Headache (Nervous system disorders) | 5 (11) | 3 (3) | 7 (10)
Pain - Joint (Musculoskeletal and connective tissue disorders) | 6 (18) | 1 (1) | 4 (5)
Pain - Muscle (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (2) | 2 (4)
Pain - Pain Nos (General disorders) | 7 (10) | 3 (3) | 5 (5)
Palpitations (Cardiac disorders) | 2 (3) | 0 (0) | 0 (0)
Platelets (Investigations) | 9 (22) | 2 (3) | 16 (47)
Pleural Effusion (Non-Malignant) (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 3 (7)
Pruritus/Itching (Skin and subcutaneous tissue disorders) | 1 (3) | 5 (5) | 6 (14)
Pulmonary/Upper Respiratory - Other (Specify, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3) | 1 (2) — Pneumonia/sinusitis/sinus congestion/nasal drainage
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 1 (5) | 9 (11) | 7 (9)
Rash: Acne/Acneiform (Skin and subcutaneous tissue disorders) | 11 (17) | 22 (30) | 24 (35)
Rash: Hand-Foot Skin Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (5) | 2 (3)
Taste Alteration (Dysgeusia) (Nervous system disorders) | 3 (4) | 4 (4) | 3 (4)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 1 (1) | 0 (0) | 5 (5)
Vision-Blurred Vision (Eye disorders) | 4 (4) | 1 (5) | 2 (3)
Vomiting (Gastrointestinal disorders) | 6 (11) | 2 (2) | 5 (8)
Weight Loss (Investigations) | 8 (10) | 6 (10) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes